CLINICAL TRIAL: NCT03172208
Title: A Phase I Single Center, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Caplacizumab in Japanese and White Healthy Volunteers.
Brief Title: Caplacizumab Single and Multiple Dose Study in Healthy Japanese and White Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ALX0681-C103
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Group 1: Japanese - Caplacizumab Dose 1 iv (SD) (Experimental): Single dose (SD) of Caplacizumab Dose 1 administered intravenously (iv) to Japanese participants
  Interventions: Biological: Caplacizumab Dose 1 iv (single-dose)
- Group 1: Japanese - Placebo iv (SD) (Placebo Comparator): Single dose (SD) of Placebo administered intravenously (iv) to Japanese participants
  Interventions: Other: Placebo iv (single-dose)
- Group 2: Japanese - Caplacizumab Dose 2 iv (SD) (Experimental): Single dose (SD) of Caplacizumab Dose 2 administered intravenously (iv) to Japanese participants
  Interventions: Biological: Caplacizumab Dose 2 iv (single-dose)
- Group 2: Japanese - Placebo iv (SD) (Experimental): Single dose (SD) of Placebo administered intravenously (iv) to Japanese participants
  Interventions: Other: Placebo iv (single-dose)
- Group 2: White - Caplacizumab Dose 2 iv (SD) (Experimental): Single dose (SD) of Caplacizumab Dose 2 administered intravenously (iv) to White participants
  Interventions: Biological: Caplacizumab Dose 2 iv (single-dose)
- Group 2: White - Placebo iv (SD) (Placebo Comparator): Single dose (SD) of Placebo administered intravenously (iv) to White participants
  Interventions: Other: Placebo iv (single-dose)
- Group 3: Japanese - Caplacizumab Dose 2 sc (SD) (Experimental): Single dose (SD) of Caplacizumab Dose 2 administered subcutaneously (sc) to Japanese participants
  Interventions: Biological: Caplacizumab Dose 2 sc (single-dose)
- Group 3: Japanese - Placebo sc (SD) (Placebo Comparator): Single dose (SD) of Placebo administered subcutaneously (sc) to Japanese participants
  Interventions: Other: Placebo sc (single-dose)
- Group 3: White - Caplacizumab Dose 2 sc (SD) (Experimental): Single dose (SD) of Caplacizumab Dose 2 administered subcutaneously (sc) to White participants
  Interventions: Biological: Caplacizumab Dose 2 sc (single-dose)
- Group 3: White - Placebo sc (SD) (Placebo Comparator): Single dose (SD) Placebo administered subcutaneously (sc) to White participants
  Interventions: Other: Placebo sc (single-dose)
- Group 4: Japanese - Caplacizumab Dose 2 sc (MD) (Experimental): Multiple doses (MD) of Caplacizumab Dose 2 administered subcutaneously (sc) to Japanese participants
  Interventions: Biological: Caplacizumab Dose 2 sc (multiple-dose)
- Group 4: Japanese - Placebo sc (MD) (Placebo Comparator): Multiple doses (MD) of Placebo administered subcutaneously (sc) to Japanese participants
  Interventions: Other: Placebo sc (multiple-dose)

INTERVENTIONS:
Biological: Caplacizumab Dose 1 iv (single-dose) — Single intravenous (iv) administration of Caplacizumab Dose 1
  Arms: Group 1: Japanese - Caplacizumab Dose 1 iv (SD)
Biological: Caplacizumab Dose 2 iv (single-dose) — Single intravenous (iv) administration of Caplacizumab Dose 2
  Arms: Group 2: Japanese - Caplacizumab Dose 2 iv (SD); Group 2: White - Caplacizumab Dose 2 iv (SD)
Biological: Caplacizumab Dose 2 sc (single-dose) — Single subcutaneous (sc) administration of Caplacizumab Dose 2
  Arms: Group 3: Japanese - Caplacizumab Dose 2 sc (SD); Group 3: White - Caplacizumab Dose 2 sc (SD)
Biological: Caplacizumab Dose 2 sc (multiple-dose) — Once daily subcutaneous (sc) administration of Caplacizumab Dose 2 during 7 consecutive days
  Arms: Group 4: Japanese - Caplacizumab Dose 2 sc (MD)
Other: Placebo iv (single-dose) — Single intravenous (iv) administration of Placebo
  Arms: Group 1: Japanese - Placebo iv (SD); Group 2: Japanese - Placebo iv (SD); Group 2: White - Placebo iv (SD)
Other: Placebo sc (single-dose) — Single subcutaneous (sc) administration of Placebo
  Arms: Group 3: Japanese - Placebo sc (SD); Group 3: White - Placebo sc (SD)
Other: Placebo sc (multiple-dose) — Once daily subcutaneous (sc) administration of Placebo during 7 consecutive days
  Arms: Group 4: Japanese - Placebo sc (MD)

SUMMARY:
Primary objective:

To assess the safety and tolerability of single ascending intravenous (i.v.) doses, a single subcutaneous (s.c.) dose of caplacizumab (Part I), and multiple s.c. doses of caplacizumab (Part II) in Japanese subjects.

Secondary objectives:

* To compare the pharmacokinetic (PK) and pharmacodynamic (PD) profiles (total vWF:Ag concentration levels [vWF:Ag], coagulation factor VIII [FVIII:C], and ristocetin cofactor activity [RICO]) after single i.v. or s.c. administration of caplacizumab in Japanese and White subjects.
* To evaluate the immunogenicity of caplacizumab (anti-drug antibodies [ADA]) in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between ≥18 kg/m² and <30 kg/m² at time of screening
* Body weight between ≥45 kg and <100 kg
* Baseline vWF:Ag between ≥60% and <170% (0.6-1.7 IU/mL)

Exclusion Criteria:

* History of and/or any sign or symptom indicating current abnormal hemostasis or blood dyscrasia, including but not limited to thrombocytopenia, thrombocytopathy, thromboasthenia, hemophilia, von Willebrand's disease, vascular purpura, bleeding gums and/or frequent nose bleeding, easy/spontaneous bruises, meno- or metrorrhagia, history of gastrointestinal bleeding or excessive bleeding after minor injury such as shaving.
* Family history of congenital vascular malformation (e.g., Marfan's Syndrome) and/or bleeding disorder (e.g., hemophilia, von Willebrand's disease, Christmas disease)
* Any surgical intervention (including tooth extraction) or trauma within the 4 weeks preceding screening for the study or any planned surgical intervention during the participation in the study
* Treatment with vitamin K, direct oral anticoagulant (DOAC), warfarin, high dose heparin within 2 weeks before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
The number of treatment-emergent adverse events (Safety and Tolerability) | From signing of informed consent form until Day 28 (single-dose part) or Day 34 (multiple dose part)

SECONDARY OUTCOMES:
Pharmacokinetics: concentration of caplacizumab in plasma | From Day -1 to Day 6 (single dose part) or to Day 12 (multiple dose part)
Pharmacokinetics: concentration of caplacizumab in urine | From Day 1 to Day 4 (single dose part) or to Day 8 (multiple dose part)
Pharmacodynamics as measured by Ristocetin cofactor activity in plasma | From Day -1 to Day 6 (single dose part) or to Day 12 (multiple dose part)
Pharmacodynamics as measured by von Willebrand factor antigen in plasma | From screening to Day 6 (single dose part) or to Day 12 (multiple dose part)
Pharmacodynamics as measured by Factor VIII clotting activity in plasma | From Day -1 to Day 6 (single dose part) or to Day 12 (multiple dose part)
Immunogenicity as measured by the concentration of anti-caplacizumab antibodies in serum | From screening until Day 28 (single-dose part) or Day 34 (multiple dose part)

CONTACTS AND LOCATIONS:
Overall Officials: Ablynx Clinical Department, Study Director — Ablynx, a Sanofi company
Locations (1):
- Investigator Site, Glendale, California, United States